CLINICAL TRIAL: NCT04126044
Title: A DOUBLE BLIND, RANDOMIZED, PARALLEL-GROUP, SINGLE-DOSE, 2-ARM, COMPARATIVE PHARMACOKINETIC STUDY OF PF-06439535 (CN) AND BEVACIZUMAB SOURCED FROM EUROPEAN UNION ADMINISTERED TO CHINESE HEALTHY MALE VOLUNTEERS
Brief Title: A SINGLE-DOSE, 2-ARM, PHARMACOKINETIC STUDY OF PF-06439535 (CN) AND EUROPEAN UNION SOURCED BEVACIZUMAB IN CHINESE HEALTHY MALE VOLUNTEERS
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was withdrawn prior to enrollment after a comprehensive review of the biosimilars market and the company's global manufacturing network.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B7391005
Record Dates: First submitted 2019-09-26; First posted 2019-10-14 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Pharmacokinetics
Keywords: Pharmacokinetics
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference: bevacizumab - EU (Active Comparator)
  Interventions: Drug: bevacizumab - EU
- Test: PF-06439535 (CN) (Experimental)
  Interventions: Drug: PF-06439535 (CN)

INTERVENTIONS:
Drug: PF-06439535 (CN) — This is the test drug Pfizer biosimilar of bevacizumab-EU.
  Arms: Test: PF-06439535 (CN)
Drug: bevacizumab - EU — This is the reference drug bevacizumab sourced from EU
  Arms: Reference: bevacizumab - EU

SUMMARY:
This is a double-blind, randomized (1:1), parallel group, single dose, 2-arm, comparative PK study of PF-06439535 (CN) and bevacizumab-EU administered intravenously to Chinese healthy male volunteers. Approximately 66 subjects will be enrolled to ensure that at least 58 subjects (29 per arm) complete the study procedures and have evaluable PK data. The study will be conducted at 1 center in China.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Chinese male subjects who, at the time of screening, are between the ages of 21 55 years of age, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate (PR) measurement, 12 lead electrocardiogram (ECG), or clinical laboratory tests.
2. Subjects must have adequate organ function (excluding subjects who received blood transfusions) according to the following laboratory values: bone marrow function (absolute neutrophil count (ANC) >=1,500/mm3 and platelet count of 100,000/mm3), adequate liver function (alanine aminotransferase (ALT) <=3 times upper limit normal and alkaline phosphatase <= 2 times upper limit normal, total bilirubin <= 1.5 mg/dl), and adequate renal function (blood urea nitrogen (BUN)/urea <=1.5 times institutional normal and Creatinine <1.5 mg/dl) upon study entry.
3. Body Mass Index (BMI) of 18 to 28 kg/m2; and a total body weight >50 kg (110 lbs).
4. Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
5. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. Evidence or history of heart failure, arterial or venous thromboembolism, bleeding diathesis, acquired coagulopathy or coagulopathy factor abnormality with international normalized ratio (INR) of >=1.5, or history of gross hemorrhage within the past 6 months prior to Screening (eg, hemoptysis or hematuria requiring medical intervention).
3. Evidence or history of relevant and clinically significant intra abdominal inflammation, gastrointestinal perforation or gall bladder perforation.
4. Major surgery or elective surgery within 3 months before or after administration of study treatment. At least 28 days should elapse from the time of minor surgical procedure, including placement of an access device and dental procedures.
5. Wounds that have not completely healed, active ulcer(s), or bone fracture(s).
6. Previous history of cancer, except for adequately treated basal cell or squamous cell carcinoma of the skin.
7. Screening supine BP >= 140 mm Hg (systolic) or >= 90 mm Hg (diastolic) on a single measurement (confirmed by a single repeat, if necessary) following at least 5 minutes of rest. If BP is >= 140 mm Hg (systolic) or >= 90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the subject's eligibility.
8. Clinically significant abnormalities in laboratory test results.
9. Screening supine 12 lead ECG demonstrating a corrected QT (QTc) interval >450 msec or a QRS interval >120 msec. If QTc exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated 2 more times and the average of the 3 QTc or QRS values should be used to determine the subject's eligibility.
10. Fertile male subjects who are unwilling or unable to use highly effective methods of contraception as outlined in this protocol (refer to Section 4.4.4) for 71 days following study drug administration.
11. A positive urine drug test.
12. History of febrile illness within 5 days prior to dosing.
13. Current use of tobacco or nicotine containing products in excess of the equivalent of 5 cigarettes per day.
14. History of regular alcohol consumption exceeding 14 drinks/week (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of Screening.
15. History of serious allergic or anaphylactic reaction to a therapeutic drug.
16. Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of investigational product (whichever is longer).
17. Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product. Use of anti platelet therapy eg, non steroidal anti inflammatory drugs (NSAIDs) is excluded. Herbal supplements must be discontinued 28 days prior to the first dose of investigational product. As an exception, acetaminophen/paracetamol may be used at doses of <=1 g/day. Limited use of non prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case by case basis, following approval by the sponsor.
18. Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
19. History of sensitivity to heparin or heparin induced thrombocytopenia.
20. Unwilling or unable to comply with the criteria in the Lifestyle Requirements section of this protocol.
21. History of human immunodeficiency virus (HIV), hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), hepatitis B core antibody (HepBcAb), or hepatitis C antibody (HCVAb).
22. Subjects who are investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees, including their family members, directly involved in the conduct of the study.
23. Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2021-01-22 (Estimated); Primary Completion 2021-07-10 (Estimated); Study Completion 2021-07-10 (Estimated)

PRIMARY OUTCOMES:
AUC0-t (Area under the serum concentration-time profile from time 0 to last time point with quantifiable concentration) | From Day 1 to Day 71

SECONDARY OUTCOMES:
Cmax (Maximum observed concentration derived from serum) | From Day 1 to Day 71
AUCinf (Area under the serum concentration-time profile from time zero extrapolated to infinity) | From Day 1 to Day 71
terminal half-life (t1/2) | From Day 1 to Day 71
clerance (CL) | From Day 1 to Day 71
steady state volume of distribution (Vss) | From Day 1 to Day 71
Percentage of participants with treatment emergent adverse events | From screening until Day 71 (total period of approximately 99 days)
Percentage of participants with clinical laboratory test results above/below certain threshold | At screening; Days -1, 2, 8, 29, 71
Incidence of anti-drug antibodies (ADA) | From day 1 to day 71
Incidence of neutralizing antibodies (Nab) | From Day 1 to Day 71

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Huashan Hospital,Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7391005